CLINICAL TRIAL: NCT00908414
Title: Phase I, Double-blind, Randomized, Placebo-controlled Trial in Healthy Volunteers to Examine Safety, Tolerability, Plasma Pharmacokinetics of TMC589337&TMC589354 After Increasing Single Oral Doses & in an Open-label Part After Different Repeated Doses in Combination With Single Oral Dose of TMC310911
Brief Title: PEPI-TiDP23-C104 is a First in Human Study With a Single Dose Escalation Part and a Multiple Dosing Part for Compounds TMC589337 and TMC589354.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: strategic decision
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR016195; PEPI-TIDP23-C104 (Other: Tibotec Pharmaceuticals Limited, Ireland)
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: HIV Infections
Keywords: PEPI-TiDP23-C104; PEPI-C104; PEPI; TMC589337; TMC589354; TMC310911; Healthy Volunteers
MeSH Terms: conditions — HIV Infections | interventions — TMC-310911

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (7):
- Panel 1: Single Dose Escalation (Experimental): Panel 1 will receive doses of 40 milligram (mg) (Session Ia), 100 mg (Session IIa), 200 mg (Session IIIa) and 400 mg (Session IVa) of TMC589337 or placebo.
  Interventions: Drug: TMC589337 40 mg; Drug: TMC589337 100 mg; Drug: TMC589337 200 mg; Drug: TMC589337 400 mg; Drug: Placebo
- Panel 2: Single Dose Escalation (Experimental): Panel 2 will receive doses of 40 mg (Session Ib), 100 mg (Session IIb), 200 mg (Session IIIb) and 400 mg (Session IVb) of TMC589354 or placebo.
  Interventions: Drug: TMC589354 40 mg; Drug: TMC589354 100 mg; Drug: TMC589354 200 mg; Drug: TMC589354 400 mg; Drug: Placebo
- Panel 3: Multiple dosing (Experimental): AA mg (Final doses will be selected based upon data obtained in the single dose sessions (i.e., Sessions I, II, and III) TMC589337 (n=6) b.i.d. (twice daily) during 7 days (Session Va) plus a single oral dose of 300 mg of TMC310911 on Day 7. After at least 14 days following Day 7 of multiple dosing, participants will receive 300 mg TMC310911, single dose (Session VIIIa).
  Interventions: Drug: TMC589337 AA mg; Drug: TMC310911 300 mg
- Panel 4: Multiple dosing (Experimental): BB mg (final doses will be selected based upon data obtained in the single dose sessions (i.e., Sessions I, II, and III) TMC589354 (n=6) b.i.d. during 7 days (Session Vb) ) plus a single oral dose of 300 mg of TMC310911 on Day 7. After at least 14 days following Day 7 of multiple dosing, participants will receive 300 mg TMC310911, single dose (Session VIIIb).
  Interventions: Drug: TMC589354 BB mg; Drug: TMC310911 300 mg
- Panel 5: Multiple dosing (Experimental): CC mg (final doses will be selected based upon data obtained in the single dose sessions (i.e., Sessions I, II, and III) TMC589337 (n=6) b.i.d. during 7 days (Session VIa) plus a single oral dose of 300 mg of TMC310911 on Day 7. After at least 14 days following Day 7 of multiple dosing, participants will receive 300 mg TMC310911, single dose (Session IXa).
  Interventions: Drug: TMC589337 CC mg; Drug: TMC310911 300 mg
- Panel 6: Multiple dosing (Experimental): DD mg (final doses will be selected based upon data obtained in the single dose sessions (i.e., Sessions I, II, and III) TMC589354 (n=6) b.i.d. during 7 days (Session VIb) ) plus a single oral dose of 300 mg of TMC310911 on Day 7. After at least 14 days following Day 7 of multiple dosing, participants will receive 300 mg TMC310911, single dose (Session IXb).
  Interventions: Drug: TMC589354 DD mg; Drug: TMC310911 300 mg
- Panel 7: Multiple dosing (Experimental): EE mg (final doses will be selected based upon data obtained in the single dose sessions (i.e., Sessions I, II, and III) TMC589337 (n=6) or YY mg TMC589354 (n=6) b.i.d. or q.d. during 7 days (Session VII) ) plus a single oral dose of 300 mg or 600mg of TMC310911 on Day 7. After at least 14 days following Day 7 of multiple dosing, participants will receive 300 mg or 600 mg TMC310911, single dose (Session X).
  Interventions: Drug: TMC589337 EE mg; Drug: TMC589354 YY mg; Drug: TMC310911 300 mg; Drug: TMC310911 600 mg

INTERVENTIONS:
Drug: TMC589337 40 mg — Participants will receive TMC589337 40 mg in Session Ia of Panel 1.
  Arms: Panel 1: Single Dose Escalation
Drug: TMC589337 100 mg — Participants will receive TMC589337 100 mg in Session IIa of Panel 1.
  Arms: Panel 1: Single Dose Escalation
Drug: TMC589337 200 mg — Participants will receive TMC589337 200 mg in Session IIIa of Panel 1.
  Arms: Panel 1: Single Dose Escalation
Drug: TMC589337 400 mg — Participants will receive TMC589337 400 mg in Session IVa of Panel 1.
  Arms: Panel 1: Single Dose Escalation
Drug: TMC589354 40 mg — Participants will receive TMC589354 40 mg in Session Ib of Panel 2.
  Arms: Panel 2: Single Dose Escalation
Drug: TMC589354 100 mg — Participants will receive TMC589354 100 mg in Session IIb of Panel 2.
  Arms: Panel 2: Single Dose Escalation
Drug: TMC589354 200 mg — Participants will receive TMC589354 200 mg in Session IIIb of Panel 2.
  Arms: Panel 2: Single Dose Escalation
Drug: TMC589354 400 mg — Participants will receive TMC589354 400 mg in Session IVb of Panel 2.
  Arms: Panel 2: Single Dose Escalation
Drug: TMC589337 AA mg — Participants will receive TMC589337 AA mg on Days 1 to 7 in Session Va of Panel 3.
  Arms: Panel 3: Multiple dosing
Drug: TMC589354 BB mg — Participants will receive TMC589354 BB mg on Days 1 to 7 in Session Vb of Panel 4.
  Arms: Panel 4: Multiple dosing
Drug: TMC589337 CC mg — Participants will receive TMC589337 CC mg on Days 1 to 7 in Session VIa of Panel 5.
  Arms: Panel 5: Multiple dosing
Drug: TMC589354 DD mg — Participants will receive TMC589354 DD mg on Days 1 to 7 in Session VIb of Panel 6.
  Arms: Panel 6: Multiple dosing
Drug: TMC589337 EE mg — Participants will receive TMC589337 EE mg on Days 1 to 7 in Session VII of Panel 7.
  Arms: Panel 7: Multiple dosing
Drug: TMC589354 YY mg — Participants will receive TMC589354 YY mg on Days 1 to 7 in Session VII of Panel 7.
  Arms: Panel 7: Multiple dosing
Drug: TMC310911 300 mg — Participants will receive TMC310911 300 mg in Panel 3, 4, 5, 6 and 7.
  Arms: Panel 3: Multiple dosing; Panel 4: Multiple dosing; Panel 5: Multiple dosing; Panel 6: Multiple dosing; Panel 7: Multiple dosing
Drug: TMC310911 600 mg — Participants will receive TMC310911 600 mg in Panel 7.
  Arms: Panel 7: Multiple dosing
Drug: Placebo — Participants will receive matching placebo to TMC589337 or TMC589354 in Panel 1 and 2.
  Arms: Panel 1: Single Dose Escalation; Panel 2: Single Dose Escalation

SUMMARY:
The purpose of the study is to determine the safety, tolerability, and plasma pharmacokinetics (i.e., the levels of TMC589337 and TMC589354 circulating in your blood over time) of increasing single oral doses of TMC589337 and TMC589354 and of multiple increasing oral doses followed by a single dose of TMC310911 to assess the potential boosting effect on the latter compound. In this study 3 investigational new drugs are involved. These new investigational drugs called TMC589337 and TMC589354 (from the PEPI family) and TMC310911 are in process of development for the treatment of Human Immunodeficiency Virus-Type 1 (HIV-1). TMC589337 and TMC589354 are novel molecules with no antiviral activity to be used to enhance the pharmacokinetics profile of a drug. TMC310911 is a novel and potent compound and belongs to a medication class called protease inhibitors (PI).

DETAILED DESCRIPTION:
This is a First-in-Human Phase I, double-blind (neither physician or patient knows the name of the assigned study drug), randomized (study medication assigned by chance), placebo-controlled (a group of study participants who receive an inactive substance in place of a medication) trial to examine the safety, tolerability, and plasma pharmacokinetics (pk) after increasing single oral doses of TMC589337 and TMC589354, and in an open-label (both the physician and study participant know the name of the assigned study drug) part after different repeated oral doses in combination with a single oral dose of TMC310911 to assess the potential pharmacokinetic enhancement on the latter compound. TMC589337 and TMC589354 are molecules to be used to enhance the pharmacokinetics profile of a drug, e.g., a Human Immunodeficiency Virus-Type 1 (HIV-1) protease inhibitors (PI). TMC310911 is an investigational PI, currently studied in healthy volunteers. The trial consists of 2 parts: a single dose escalation part (double-blind, placebo-controlled) and a multiple dosing part (open label) for both PEPI-compounds: TMC589337 and TMC589354. The single dose escalation part of the trial will include 2 panels of 8 healthy adult volunteers each (Panel 1 and 2). Each panel will have 4 oral escalating single dose sessions of either TMC589337 (Panel 1) or TMC589354 (Panel 2). Healthy volunteers will receive doses of 40 mg (Session Ia), 100 mg (Session IIa), 200 mg (Session IIIa) and 400 mg (Session IVa) of TMC589337 or placebo. Panel 2 will receive doses of 40 mg (Session Ib), 100 mg (Session IIb), 200 mg (Session IIIb) and 400 mg (Session IVb) of TMC589354 or placebo. Both panels can run in parallel. In each session, 6 healthy volunteers will receive active treatment and 2 healthy volunteers will receive placebo with standard meals. Doses of 40 mg, 100 mg, 200 mg and 400 mg of TMC589337 or TMC589354 or placebo will be administered as a single oral administration. The treatment schedule will be made in such a way that for both panels over 4 sessions each healthy volunteer will receive active treatment 3 times and placebo once. A washout period (a period where no treatment will be taken in view of having all the medication eliminated from the body before starting a new treatment) of at least 10 days will be respected between consecutive TMC589337, TMC589354 or placebo dosing within each panel. Each single dosing session will have a staggered approach meaning that first 4 healthy volunteers will be dosed and 48 hours later the next 4 healthy volunteers will be dosed. Multiple dosing will be started when the 200 mg sessions of TMC589337 and/or TMC589354 are found to be generally safe and well tolerated as decided by the Investigator and the Sponsor and approved as such by the local ethics committee. Multiple dosing of TMC589337 and/or TMC589354 will not be started if the plasma pk profile is not supportive to evaluate repeated dosing. The multiple dose part of the trial is open-label and will include 5 panels of 6 healthy adult volunteers each (Panels 3, 4, 5, 6 and 7). Each panel will have 1 session in which TMC589337 or TMC589354 will be administered. Treatment is anticipated to be a twice daily regimen, and different dose regimens will be tested. Final doses will be determined according to the results obtained from the single dose sessions but will not be higher than a total daily dose of 400 mg. If multiple dosing is found to be generally safe and well tolerated in Panel 3 and 4, doses for Panels 5-7 can be determined. Both Panels 3 and 4, and Panels 5 and 6 can run in parallel. In Panel 7, 1 compound, either TMC589337 or TMC589354, will be selected for a twice daily or once daily regimen for 7 days. In addition, the healthy volunteers of Panels 3, 4, 5 and 6 will receive a single oral dose of 300 mg of TMC310911 on Day 7 of these sessions to assess the enhancing effect of repeated administration of TMC589337 and TMC589354 on the pk profile of a single dose of TMC310911. Healthy volunteers of Panel 7 will receive either a 300 mg dose of TMC310911 or a dose of 600 mg TMC310911 at the same conditions. Study medication will be given under fed conditions in Panels 3-6, and under fed or fasted conditions (depending on the findings of previous sessions) in Panel 7. After a washout period of at least 14 days healthy volunteers of Panels 3 to 7 will have an additional session in which a single oral dose of 300 mg (or 600 mg for Panel 7 only) of TMC310911 alone will be administered (Sessions VIIIa, VIIIb, IXa, IXb and X). Full pk profiles of TMC589337 and TMC589354 will be determined up to 72 hours after single dosing and after the morning dosing of Day 7 (multiple dosing), and over 12 hours (or over 24 hours for Panel 7 when given once daily.) after the morning dose on Days 1 and 6 of the multiple dosing sessions. Full pk profiles of TMC310911 will be determined over 24 hours when given alone and on Day 7 of the TMC589337 and TMC589354 multiple dosing sessions. Safety and tolerability will be evaluated continuously and documented (safety report) before stepping up to the next dose. Dose escalation in the single and multiple ascending dose regimens will continue only if the previous dose was found safe and generally well tolerated by the Investigator and the Sponsor and approved as such by the ethics committee. Actual doses may be adapted pending on the outcome of the previous sessions. The expected duration of the study (excluding screening) is at least 8 weeks. Safety and tolerability evaluations will be recorded at regular intervals throughout the trial period. Illnesses and side effects will be monitored continuously. Blood and urine samples will be taken at screening, in Panel 1 and 2 on Day 1, 2 and 4 of sessions I to IV, in Panel 3 to 7 on Day 1, 3, 6, 7, 8 and 10 of session V, VI and VII, on Day 1 and 2 of session VIII, IX and X and at the 2 follow-up visits 10 to 14 days and 30 to 32 days after last drug intake. Electrocardiogram (ECG) will be taken and vital signs (blood pressure and heart rate) will be measured at screening, in Panel 1 and 2 at each session day ( on Day -1 only ECGs), in Panel 3 to 7 at Day -1 (only ECG), Day 1, 3, 6, 7, 8 and 10 in session V, VI and VII and on Day 1 and 2 of session VIII, IX and X and at the 2 follow-up visits. Physical examination will be done at screening, on Day 4 of each session in Panel 1 and 2, on Day 6 and 10 of session V, VI and VII, on Day -1 and 2 of session VIII, IX and X and at the 2 follow-up visits. Continuous ECG data will be obtained during the first 8 hours after intake of study medication in the single dose escalation part of the study. TMC589337,TMC589354,TMC310911 and placebo are formulated as oral drinkable solutions. Panel 1-2 consist of single dose of TMC589337 or TMC589354 and placebo from 40-400mg (2ml to 5ml) on Day 1 of each session. Panel 3-7 consist of TMC589337,TMC589354 or placebo twice daily (or once daily in Panel 7), from Day 1 to Day 7 with maximum daily dose of 400mg (5ml) plus a single morning intake of 300mg (12ml) (or 600mg for Panel 7 only) TMC310911 on Day 7 and on Day 1 in 2nd session.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmokers for at least 3 months prior to selection
* Weight as defined by a Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included
* Informed Consent Form (ICF) signed voluntarily
* Able to comply with protocol requirements
* Healthy on the basis of a pretrial physical examination, medical history, the results of blood biochemistry and hematology tests, a urinalysis, vital signs, and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* Past history of clinically significant heart arrhythmias (extrasystolic, tachycardia at rest)
* having baseline prolongation of QTc interval > 450 ms, history of risk factors for Torsade de Pointes syndrome (hypokalemia, family history of long QT Syndrome)
* Female, except if postmenopausal for more than 2 years, or posthysterectomy or postsurgical sterilization (without reversal operation)
* Currently active clinically relevant or significant underlying gastrointestinal, cardiovascular, nervous system, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease
* History of clinically relevant skin disease or allergy including drug allergy as well.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
The trial objectives are to determine the safety, tolerability and plasma pk of TMC589337/TMC589354 after increasing single oral doses from 40 mg up to 400 mg and after increasing multiple oral doses. | 8 weeks. This includes a treatment, washout and follow up period and is excluding screening period of maximum 21 days before first medication intake)

SECONDARY OUTCOMES:
The trial objectives are to determine the safety, tolerability and plasma pk interaction between TMC310911 and TMC589337 or TMC589354. | 8 weeks. This includes a treatment, washout and follow up period and is excluding screening period of maximum 21 days before first medication intake)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (1):
- Utrecht, Netherlands